CLINICAL TRIAL: NCT02111681
Title: Calypso-based Deep Inspiration Breath Hold (DIBH) Radiation Treatments of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-174
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Calypso-based Deep Inspiration Breath Hold (DIBH); radiation treatments; 13-174
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- Calypso-based Deep Inspiration Breath Hold (DIBH) (Experimental): This trial will investigate the feasibility of implanted anchored Beacon ® electromagnetic lung transponders (Calypso ®) to guide and monitor deep-inspiration breathhold (DIBH) treatments in patients with inoperable thoracic malignancies.
  Bronchoscopic Calypso Beacon Implantation, Simulation - Free-breathing scan - 4D CT scan,- DIBH CT scan Radiation - Treatment setup, - Calypso signal recording, - RT treatment with DIBH with or without visual biofeedback Follow-up - 3 and 6 months after RT with diagnostic CT chest
  Interventions: Device: Calypso Beacon Implantation

INTERVENTIONS:
Device: Calypso Beacon Implantation — Bronchoscopic Calypso Beacon Implantation

SUMMARY:
The purpose of this study is to test the use of Calypso beacon implants as a way to determine where the lung tumor is located during radiation treatment. The Calypso beacons are small devices that are implanted in the lungs, near the tumor. They are able to send a signal to a tracking system to show where they are, and where the tumor is, as the patient holds their breath for the radiation treatment. The investigators want to find out what effects, good and/or bad, that this has on the patient and the way they treat the cancer in your lungs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of malignancy suitable for thoracic radiation therapy
* Patients planning to undergo radiation therapy for primary or recurrent malignancy of the lung or metastatic malignancy to the lung.
* Age ≥ 18 years old
* KPS ≥ 60%
* Ability to hold their breath for >20 seconds for 5 times
* Patients who are able to tolerate flexible bronchoscopy
* Patients with life expectancy of at least 12 months
* Patients able to have bronchoscopic placement of Calypso as confirmed on a recent (within the past 8 weeks) CT scan.
* Patients who are able to comply with the protocol follow-up schedule.

Exclusion Criteria:

* Patients unable to comply with instructions for DIBH
* Patients with implants in the chest region that contain metal or conductive materials (e.g., metal implants, rods, or plates) which Calypso Medical considers will interfere with the Calypso System's electromagnetic localization.
* Patients with active implanted devices, such as pacemakers, defibrillators, and drug infusion pumps since the effects of the Calypso System operation on these devices are unknown.
* Patients with clinically significant active infections.
* Patients with bronchiectasis in the region of the intended implantation sites.
* Patients with a history of hypersensitivity to nickel.
* Patients whose lung tumors are being monitored with MR imaging (MR imaging of the anchored transponders is safe but yields an image artifact around the anchored transponders).
* Posterior lesions that would be >19cm distance from Calypso detector plate. Patients may be treated in the prone position in order to meet the required minimum distance.
* Patients with any other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in this clinical study.
* Patients who are deemed unable to safely undergo or tolerate flexible bronchoscopy
* Patients who are unable to tolerate anesthesia or sedation
* Patients enrolled in any other clinical studies the investigator believes to be in conflict with this investigation.
* Female patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daphna Gelblum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Calypso-based Deep Inspiration Breath Hold (DIBH): This trial will investigate the feasibility of implanted anchored Beacon ® electromagnetic lung transponders (Calypso ®) to guide and monitor deep-inspiration breathhold (DIBH) treatments in patients with inoperable thoracic malignancies.
  Bronchoscopic Calypso Beacon Implantation, Simulation - Free-breathing scan - 4D CT scan,- DIBH CT scan Radiation - Treatment setup, - Calypso signal recording, - RT treatment with DIBH with or without visual biofeedback Follow-up - 3 and 6 months after RT with diagnostic CT chest
  Calypso Beacon Implantation: Bronchoscopic Calypso Beacon Implantation
Period: Overall Study
Arm/Group | Calypso-based Deep Inspiration Breath Hold (DIBH)
Started | 48
Completed | 37
Not Completed | 11
Not completed — Death | 5
Not completed — Lack of Efficacy | 2
Not completed — Progression of disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Calypso-based Deep Inspiration Breath Hold (DIBH)
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 69 [60 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Calypso Transponders
Description: Feasibility is defined as completion of all treatments using the DIBH treatment plan and Calypso transponders.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Calypso-based Deep Inspiration Breath Hold (DIBH)
Number analyzed (Participants) | 48
Participants
  Participants who completed all treatments using DIBH treatment plan and Calypso transponders | 46
  Participants who did not complete all treatments using DIBH treatment plan and Calypso transponders | 2

2. Secondary Outcome: Reproducibility
Description: We will compare the visual vs no visual biofeedback treatments (done for each patient) by the number of treatment interruptions.
Time Frame: 2 years
Population: Data not collected due to the study team being unable to secure appropriate visual feedback devices to assess this objective.
Arm/Group | Calypso-based Deep Inspiration Breath Hold (DIBH)
Number analyzed (Participants) | 0

3. Secondary Outcome: Measure the Residual Intrafraction Tumor Motion
Description: will be measured in all 3 dimensions and the euclidean distance will be calculated in milimeters/mm, which will then be correlated with the normal tissue dosimetry by regression analysis.
Time Frame: 2 years
Measure: Mean (Full Range); unit: mm
Arm/Group | Calypso-based Deep Inspiration Breath Hold (DIBH)
Number analyzed (Participants) | 48
mm | 3 [2 to 5]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Calypso-based Deep Inspiration Breath Hold (DIBH)
All-Cause Mortality (participants affected / at risk) | 30/48
Serious Adverse Events (participants affected / at risk) | 8/48
Other Adverse Events (participants affected / at risk) | 10/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calypso-based Deep Inspiration Breath Hold (DIBH) (N=48)
Esophagitis (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
IV contrast allergy (Injury, poisoning and procedural complications) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Bacteremia (Infections and infestations) | 1
Fever (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calypso-based Deep Inspiration Breath Hold (DIBH) (N=48)
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 3
Supraventricular tachycardia/SVT (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT02111681/Prot_SAP_000.pdf